CLINICAL TRIAL: NCT00989742
Title: A Randomised, Double Blind, Placebo Controlled Trial of Doxycycline in Lymphangioleiomyomatosis.
Brief Title: Doxycycline In Lymphangioleiomyomatosis (LAM)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 07061
Record Dates: First submitted 2009-10-02; First posted 2009-10-05 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Lymphangioleiomyomatosis; Tuberous Sclerosis
Keywords: lymphangioleiomatosis; LAM; tuberous sclerosis; doxycycline; matrix metalloproteinases; MMP
MeSH Terms: conditions — Lymphangioleiomyomatosis; Tuberous Sclerosis | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Doxycycline (Active Comparator)
  Interventions: Drug: Doxycycline
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Doxycycline — 50mg od
  Arms: Doxycycline
Drug: Placebo — 50mg od
  Arms: Placebo

SUMMARY:
The purpose of the study is to test if the drug doxycycline is effective in slowing the progression of lung disease in LAM. Lymphangioleiomyomatosis (LAM) is a rare lung disease which affects young women. Women with LAM develop enlarged air spaces in the lungs called cysts, caused by an excess of matrix metalloproteinases (MMPs), protein-digesting enzymes. LAM is associated with kidney tumours, called angiomyolipomas, and causes recurrent lung collapse, breathlessness and death or need for lung transplant. There is no proven treatment. Doxycycline, a commonly used antibiotic can block MMP production and a small number of patients have shown some benefit from doxycycline. The investigators will perform a study to test if doxycycline can slow the fall in lung function in patients with LAM. Forty patients who consent to participate will take doxycycline or a placebo (dummy) tablet for two years in addition to their standard treatment.

DETAILED DESCRIPTION:
Summary

We will perform a 2 year double blind, placebo controlled trial of doxycycline in 40 patients with LAM. The main endpoints will be change in FEV1, other measures of efficacy, safety and dose required to suppress MMP activity. After clinical evaluation, lung function, shuttle walk, QoL assessment, blood tests, serum and urine MMPs (termed full assessment) plus baseline chest X-ray patients will be randomised to doxycycline 50 mg od or placebo. Patients will be assessed at 2 weeks for a safety screen, every 3 months for clinical evaluation and spirometry and at 12 and 24 months for full assessment. At 3 months urine zymography will be performed to see if MMPs are present in urine at the prescribed dose. Doxycycline will be increased to 100 mg bd at three months after urine zymography has been performed. To avoid withholding treatment from those who decline rapidly, patients who, on two occasions, have either a fall from baseline FEV1 of 300 ml or fall in resting SaO2 of 3% will be assessed by an independent expert (AET). Patients receiving placebo will be given the option of doxycycline according to protocol. Those receiving doxycycline the option of continuing in the study or withdrawal. These patients and those withdrawn due to recurrent pneumothorax, increase in chylous effusion or bleeding angiomyolipoma will be included in a composite safety endpoint and analysed on an intention to treat basis. Power calculations based on retrospective cohorts(Johnson and Tattersfield 1999) show that 20 patients per group will give 80% power to detect a 70 ml/year difference in FEV1 based an assumed SD for a fall in FEV1 of 75 ml/year. The mean slope of regression lines for FEV1 and FVC, plus change DLCO, shuttle walk distance and QoL in the doxycycline and placebo groups will be compared by parametric or non-parametric analysis dependent on data, time to composite safety endpoint by Caplan-Meier analysis, complications and adverse events by Chi Square test.

1. Introduction

Lymphangioleiomyomatosis Lymphangioleiomyomatosis (LAM) is a disease of the lungs and lymphatics, which can occur sporadically or in association with tuberous sclerosis complex (TSC). The disease is rare, occurring in 1-2 / million of the population but in up to 40% of women with TSC LAM almost exclusively affects women, generally developing before the menopause. The disease is characterised by progressive pulmonary cystic change, recurrent pneumothorax, chylous pleural collections and, in most cases, progressive respiratory failure. Abdominal manifestations caused by obstruction and dilation of the axial lymphatics include lymphadenopathy, cystic lymphatic masses (lymphangioleiomyomas), chylous ascites and angiomyolipoma (a benign tumour). Survival in LAM is, 70 90% at 10 yrs, although this is highly variable since long-term survivors have been described. Diagnosis is made by a combination of clinical features and computed tomography scanning or, in cases of doubt, lung biopsy. In patients with rapidly progressive disease, hormone treatment (predominantly progesterone) has been used, although no firm evidence supports its use. Otherwise, treatment is aimed at complications including pneumothorax, chylous collections and extra-pulmonary manifestations. The only treatment for severe LAM is currently lung transplantation(Johnson 2006). Recently identification of abnormalities in the tuberous sclerosis complex (TSC) genes in sporadic and TSC associated LAM have identified dysregulation of the mTOR pathway in LAM (Carsillo, Astrinidis et al. 2000; Sato, Seyama et al. 2002) and have lead to clinical trials of mTOR inhibitors such as rapamycin in LAM and TSC. At the time of writing these have not been reported but appear promising.

Background and preliminary data Cystic lung destruction is the hallmark of pulmonary LAM and generally results in respiratory failure over a variable period of time(Johnson 2006). Over-activity of proteases including elastase, trypsin and the matrix metalloproteinases (MMPs) is responsible for parenchymal destruction in emphysema and other lung diseases. The MMPs are a family of zinc dependent proteolytic enzymes with proteolytic activities against extra-cellular matrix proteins. The MMPs are overexpressed in inflammatory and neoplastic diseases where in addition to processing extra-cellular matrix they also have roles in metastasis, angiogenesis, growth factor activation and inactivation(Stamenkovic 2003). MMPs -1, -2, and -9 are involved in the sequential digestion of collagen and gelatin and are strongly expressed in the walls of cysts where it is thought they contribute to parenchymal destruction in LAM(Matsui, Takeda et al. 2000). Further, MMPs can be detected by gelatin zymography in the urine of patients with LAM but not controls. Doxycycline is a tetracycline antibiotic in common clinical use. In addition to its antimicrobial action it inhibits the synthesis and activity of several MMPs and inhibits proliferation of a range of cell types including arterial smooth muscle, cancer cells and cancer model systems(Bendeck, Conte et al. 2002; Duivenvoorden, Popovic et al. 2002; Onoda, Ono et al. 2004). In preliminary experiments we have demonstrated that primary LAM derived and angiomyolipoma cells produce MMP-2 and -7 and that MMP expression and proliferation in these cells in inhibited by doxycycline.

Preliminary clinical data of doxycycline in LAM In a preliminary open label study of doxycycline (50 - 100 mg qds) in 10 patients with LAM, doxycycline improved 6 minute walk distance) and Borg dyspnoea score (Glassberg et al. Data presented at the LAM Foundation International Research Conference, Cincinnati Ohio 2006). In a single case report, Moses et al. observed an improvement in FEV1 and oxygenation during exercise in a patient with LAM treated with 100mg doxycycline daily (Moses, Harper et al. 2006). In both of these cases MMP-2 and -9 were initially present in the patient's urine and was undetectable after treatment with doxycycline. In a study of 14 patients, doxycycline 100mg bd is known to give a mean plasma concentration of 4.41 µg/ml (range 1.9-9.4 µg/ml)(Prall, Longo et al. 2002).

Specific issues in orphan disease clinical trials and rationale for trial design Studying orphan diseases presents specific challenges, specifically the limited number of patients available, wide geographic distribution and low priority for funding due to the perceived poor economic benefit. Patients are well informed about potential developments due to patient groups and internet based information(Tattersfield and Glassberg 2006) and may obtain potential treatments 'off label' making definitive research studies impossible. As LAM is rare, cohorts drawn from a wide area are required for studies to achieve adequate power. We have 15 years experience of LAM research and from our UK LAM database estimate there are approximately 120 patients in the UK. We are currently performing an open label study of Sirolimus in LAM and tuberous sclerosis (TESSTAL, a Study of The Efficacy and Safety of Sirolimus (Rapamycin) Therapy for Renal Angiomyolipomas in Patients with Tuberous Sclerosis Complex And Sporadic Lymhangioleiomyomatosis). This included six patients with LAM whom we found to be well motivated and will travel long distances for study visits (including Cornwall, Kent and Perth). Despite the known adverse effects of rapamycin six of eight eligible (i.e. with LAM and angiomyolipoma) patients invited took part in the study. The current study protocol has been designed as a simple protocol which is both inclusive of most patients with LAM and has a follow up which is similar to routine clinical care which we hope will facilitate recruitment. In addition the protocol is less demanding than that of the TESSTAL study. As most patients are known to us via our database or clinical contacts we expect recruitment to be complete within six months.

Designing a definitive study is difficult without having an estimate of the likely size of effect, if this is large, as suggested by the one case report(Moses, Harper et al. 2006) a small number of patients are needed. If it is small as seems more likely a priori, a larger number of patients are needed requiring European collaboration and considerably greater funding. We therefore designed a pragmatic pilot study using a single geographic population with a simple, inexpensive protocol which will serve several functions, specifically to: (1) determine the optimum dose of doxycycline needed to suppress MMP production. (2) define the safety profile of doxycycline in LAM. (3) provide evidence of efficacy and size of effect. (4) provide data to help optimise the design and logistics of future trials.

2 Study aims/objectives

Hypothesis Doxycycline will prevent matrix metalloproteinase dependent tissue destruction in lymphangioleiomyomatosis (LAM) thus preserving lung function, exercise capacity and quality of life.

We will perform a randomised placebo controlled trial of doxycycline on rate of decline of FEV1 over two years against matched placebo. This study will:

1. determine the optimum dose of doxycycline needed to suppress MMP production.
2. define the safety profile of doxycycline in LAM.
3. provide evidence for efficacy and size of effect.
4. provide data to help optimise the design and logistics of future trials.

With the data obtained we will be in a strong position to apply for European funding for a European wide trial should this still be required.

3 Investigational plan

Patient population and recruitment

Forty patients with either sporadic LAM or TSC-LAM will be recruited from the UK LAM database, physician referrals, LAM Action (a patients group for women with LAM) and the Tuberous Sclerosis Association. Patients will be contacted by mail by the principal investigator. Potential participants will receive a preliminary information sheet and response sheet for return by prepaid post. Those that express a potential interest in participating will be offered a face to face interview with one of the study doctors to assess eligibility, answer questions, obtain details of all physicians involved in their care and obtain written consent prior to enrolment. We anticipate recruitment will be complete within 12 months of starting the study.

ELIGIBILITY:
Inclusion Criteria:

* Sporadic LAM diagnosed either by cystic lung disease on HRCT classical of LAM plus angiomyolipoma or chylous effusion or cystic lung disease on HRCT and tissue biopsy showing LAM or angiomyolipoma
* TSC-LAM diagnosed by cystic lung disease on HRCT and tuberous sclerosis diagnosed by TSC consensus criteria(13).
* Patients with either an FEV1 below 80% predicted or evidence of a 20% deterioration in FEV1.
* Hormone and bronchodilator treatment for LAM* is allowed providing treatment has not changed in the three months prior to enrollment.

  * progesterone, GnRh agonists and bronchodilators

Exclusion Criteria:

* Inability to give informed consent.
* Mental retardation.
* Age less than 18 years.
* Pneumothorax, chylous effusion, bleeding angiomyolipoma or change in hormone treatment within 3 months.
* Previous organ transplantation.
* Severe or uncontrolled epilepsy.
* Use of any oral contraceptive pill.
* Pregnancy or breast feeding. Pre-menopausal patients must be willing to use appropriate birth control measures to avoid pregnancy while enrolled in the study.
* Major systemic diseases (malignancy, myocardial infarction or unstable angina, type1 diabetes, severe hypertension, liver cirrhosis).
* Use of drugs known to interact with doxycycline, including anticoagulation with warfarin.
* Anticoagulation with warfarin.
* Hypersensitivity to tetracyclines.
* Treatment with mTOR inhibitor within the previous 3 months (sirolimus, everolimus).
* Use of doxycycline or other experimental drug within the previous three months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Mean rate of change of FEV1 over 24 months on doxycycline compared with placebo. | 2 years

SECONDARY OUTCOMES:
Rate change FVC over 24 months Change DLCO at 12 & 24 mths Change in shuttle walk distance at 12 & 24 mths Change in QOL at 12 & 24 mths Time to composite safety endpoint Number complications Number respiratory infections Adverse effects | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Simon R Johnson, DM FRCP, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham University Hospitals, Nottingham, Nottingham, United Kingdom

REFERENCES:
- [Background] Johnson SR, Tattersfield AE. Decline in lung function in lymphangioleiomyomatosis: relation to menopause and progesterone treatment. Am J Respir Crit Care Med. 1999 Aug;160(2):628-33. doi: 10.1164/ajrccm.160.2.9901027. PMID 10430739
- [Background] Johnson SR. Lymphangioleiomyomatosis. Eur Respir J. 2006 May;27(5):1056-65. doi: 10.1183/09031936.06.00113303. PMID 16707400
- [Background] Carsillo T, Astrinidis A, Henske EP. Mutations in the tuberous sclerosis complex gene TSC2 are a cause of sporadic pulmonary lymphangioleiomyomatosis. Proc Natl Acad Sci U S A. 2000 May 23;97(11):6085-90. doi: 10.1073/pnas.97.11.6085. PMID 10823953
- [Background] Sato T, Seyama K, Fujii H, Maruyama H, Setoguchi Y, Iwakami S, Fukuchi Y, Hino O. Mutation analysis of the TSC1 and TSC2 genes in Japanese patients with pulmonary lymphangioleiomyomatosis. J Hum Genet. 2002;47(1):20-8. doi: 10.1007/s10038-002-8651-8. PMID 11829138
- [Background] Stamenkovic I. Extracellular matrix remodelling: the role of matrix metalloproteinases. J Pathol. 2003 Jul;200(4):448-64. doi: 10.1002/path.1400. PMID 12845612
- [Background] Matsui K, Takeda K, Yu ZX, Travis WD, Moss J, Ferrans VJ. Role for activation of matrix metalloproteinases in the pathogenesis of pulmonary lymphangioleiomyomatosis. Arch Pathol Lab Med. 2000 Feb;124(2):267-75. doi: 10.5858/2000-124-0267-RFAOMM. PMID 10656737
- [Background] Bendeck MP, Conte M, Zhang M, Nili N, Strauss BH, Farwell SM. Doxycycline modulates smooth muscle cell growth, migration, and matrix remodeling after arterial injury. Am J Pathol. 2002 Mar;160(3):1089-95. doi: 10.1016/S0002-9440(10)64929-2. PMID 11891205
- [Background] Onoda T, Ono T, Dhar DK, Yamanoi A, Fujii T, Nagasue N. Doxycycline inhibits cell proliferation and invasive potential: combination therapy with cyclooxygenase-2 inhibitor in human colorectal cancer cells. J Lab Clin Med. 2004 Apr;143(4):207-16. doi: 10.1016/j.lab.2003.12.012. PMID 15085079
- [Background] Duivenvoorden WC, Popovic SV, Lhotak S, Seidlitz E, Hirte HW, Tozer RG, Singh G. Doxycycline decreases tumor burden in a bone metastasis model of human breast cancer. Cancer Res. 2002 Mar 15;62(6):1588-91. PMID 11912125
- [Background] Prall AK, Longo GM, Mayhan WG, Waltke EA, Fleckten B, Thompson RW, Baxter BT. Doxycycline in patients with abdominal aortic aneurysms and in mice: comparison of serum levels and effect on aneurysm growth in mice. J Vasc Surg. 2002 May;35(5):923-9. doi: 10.1067/mva.2002.123757. PMID 12021708
- [Background] Moses MA, Harper J, Folkman J. Doxycycline treatment for lymphangioleiomyomatosis with urinary monitoring for MMPs. N Engl J Med. 2006 Jun 15;354(24):2621-2. doi: 10.1056/NEJMc053410. No abstract available. PMID 16775248
- [Background] Tattersfield AE, Glassberg MK. Lymphangioleiomyomatosis: a national registry for a rare disease. Am J Respir Crit Care Med. 2006 Jan 1;173(1):2-4. doi: 10.1164/rccm.2509010. No abstract available. PMID 16368790
- [Background] Roach ES, Gomez MR, Northrup H. Tuberous sclerosis complex consensus conference: revised clinical diagnostic criteria. J Child Neurol. 1998 Dec;13(12):624-8. doi: 10.1177/088307389801301206. PMID 9881533
- [Background] Lazor R, Valeyre D, Lacronique J, Wallaert B, Urban T, Cordier JF; Groupe d'Etudes et de Recherche sur les Maladies "Orphelines" Pulmonaires. Low initial KCO predicts rapid FEV1 decline in pulmonary lymphangioleiomyomatosis. Respir Med. 2004 Jun;98(6):536-41. doi: 10.1016/j.rmed.2003.11.013. PMID 15191039
- [Background] Taveira-DaSilva AM, Stylianou MP, Hedin CJ, Hathaway O, Moss J. Decline in lung function in patients with lymphangioleiomyomatosis treated with or without progesterone. Chest. 2004 Dec;126(6):1867-74. doi: 10.1378/chest.126.6.1867. PMID 15596686
- [Background] Johnson S, Knox A. Autocrine production of matrix metalloproteinase-2 is required for human airway smooth muscle proliferation. Am J Physiol. 1999 Dec;277(6):L1109-17. doi: 10.1152/ajplung.1999.277.6.L1109. PMID 10600880
- [Background] Henderson N, Markwick LJ, Elshaw SR, Freyer AM, Knox AJ, Johnson SR. Collagen I and thrombin activate MMP-2 by MMP-14-dependent and -independent pathways: implications for airway smooth muscle migration. Am J Physiol Lung Cell Mol Physiol. 2007 Apr;292(4):L1030-8. doi: 10.1152/ajplung.00317.2006. Epub 2006 Dec 22. PMID 17189319
- [Background] Elshaw SR, Henderson N, Knox AJ, Watson SA, Buttle DJ, Johnson SR. Matrix metalloproteinase expression and activity in human airway smooth muscle cells. Br J Pharmacol. 2004 Aug;142(8):1318-24. doi: 10.1038/sj.bjp.0705883. Epub 2004 Jul 20. PMID 15265805
- [Background] Crooks DM, Pacheco-Rodriguez G, DeCastro RM, McCoy JP Jr, Wang JA, Kumaki F, Darling T, Moss J. Molecular and genetic analysis of disseminated neoplastic cells in lymphangioleiomyomatosis. Proc Natl Acad Sci U S A. 2004 Dec 14;101(50):17462-7. doi: 10.1073/pnas.0407971101. Epub 2004 Dec 6. PMID 15583138